CLINICAL TRIAL: NCT00376025
Title: Study of the Effects of Antioxidant Supplementation in Patients Suffering From Kashin-Beck Disease
Brief Title: Antioxidant Supplementation in Patients With Kashin-Beck Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovative Humanitarian Solutions (Other)
Collaborators: University of Houston - Victoria (Other)
Responsible Party: Richard S. Gunasekera, Ph.D., Study Chair and P.I., University of Houston - Victoria
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: KB001
Record Dates: First submitted 2006-09-12; First posted 2006-09-14 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2008-02

CONDITIONS: Kashin-Beck Disease
Keywords: Kashin-Beck Disease; Kashin-Beck Osteoarthropathy
MeSH Terms: conditions — Kashin-Beck Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Biological Antioxidant Supplementation — Supplementation of affected population with the Phytochemical antioxidant, Garcinia Mangostata in addition to sodium selenate.

SUMMARY:
The purpose of this study is to determine whether antioxidant supplementation can have a positive health effect on patients suffering from Kashin-Beck disease.

DETAILED DESCRIPTION:
Current research regarding Kashin-Beck disease, (KBD) have identified dramatic deficiencies of both selenium and iodine in patients with this disease. Initial supplementation of these trace minerals provided no measurable benefit to the affected population. Research conducted by Innovative Humanitarian Solutions, suggests that such deficiencies may not be causal, but markers of an underlying condition of extreme oxidative stress brought on by the improper functioning of the Glutathione Peroxidase enzyme in synthesizing H202 during periods of critical cellular development, primarily in mesenchymal cell development.

The purpose of this trial is to determine the efficacy of antioxidant supplementation in aiding the Glutathione Peroxidase enzyme in its proper function and thereby reducing oxidative stress and enabling the uptake of selenium and iodine which are necessary for proper bone growth and development.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed patients with Kashin-Beck disease

Exclusion Criteria:

* less than 24 hours from admission to ICU
* Patients who are moribund
* Lack of commitment to program
* Absolute contraindication to enteral nutrients
* Severe acquired brain injury
* Pregnant or lactating patients
* Previous randomization in this study
* Enrollment in a related interventional study
* Child's class C liver disease Metastatic cancer with life expectancy < 6 months Seizure disorder requiring anticonvulsant medication

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-01 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Score on FLACC or Word Graphic pain rating scale at 3, 6, 9 months | One Year

SECONDARY OUTCOMES:
Increase in serum selenium concentrations at 6 months | Six Months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gunasekera, Ph.D., Study Chair — University of Houston - Victoria; Jeff C Cokenour, B.S., Principal Investigator — Innovative Humanitarian Solutions; Minh Han, M.D., Principal Investigator — Innovative Humanitarian Solutions
Locations (1):
- Lhasa Prefecture and surrounding villages, Lhasa, Tibet, China

REFERENCES:
- [Background] Moreno-Reyes R, Egrise D, Boelaert M, Goldman S, Meuris S. Iodine deficiency mitigates growth retardation and osteopenia in selenium-deficient rats. J Nutr. 2006 Mar;136(3):595-600. doi: 10.1093/jn/136.3.595. PMID 16484530
- [Background] Kohrle J, Jakob F, Contempre B, Dumont JE. Selenium, the thyroid, and the endocrine system. Endocr Rev. 2005 Dec;26(7):944-84. doi: 10.1210/er.2001-0034. Epub 2005 Sep 20. PMID 16174820
- [Background] Xia Y, Hill KE, Byrne DW, Xu J, Burk RF. Effectiveness of selenium supplements in a low-selenium area of China. Am J Clin Nutr. 2005 Apr;81(4):829-34. doi: 10.1093/ajcn/81.4.829. PMID 15817859
- [Background] Esworthy RS, Yang L, Frankel PH, Chu FF. Epithelium-specific glutathione peroxidase, Gpx2, is involved in the prevention of intestinal inflammation in selenium-deficient mice. J Nutr. 2005 Apr;135(4):740-5. doi: 10.1093/jn/135.4.740. PMID 15795427
- [Background] Beckett GJ, Arthur JR. Selenium and endocrine systems. J Endocrinol. 2005 Mar;184(3):455-65. doi: 10.1677/joe.1.05971. PMID 15749805
- [Background] Moreno-Reyes R, Mathieu F, Boelaert M, Begaux F, Suetens C, Rivera MT, Neve J, Perlmutter N, Vanderpas J. Selenium and iodine supplementation of rural Tibetan children affected by Kashin-Beck osteoarthropathy. Am J Clin Nutr. 2003 Jul;78(1):137-44. doi: 10.1093/ajcn/78.1.137. PMID 12816783
- [Background] Stamler J, Stamler R, Neaton JD, Wentworth D, Daviglus ML, Garside D, Dyer AR, Liu K, Greenland P. Low risk-factor profile and long-term cardiovascular and noncardiovascular mortality and life expectancy: findings for 5 large cohorts of young adult and middle-aged men and women. JAMA. 1999 Dec 1;282(21):2012-8. doi: 10.1001/jama.282.21.2012. PMID 10591383
- [Background] Harris NS, Crawford PB, Yangzom Y, Pinzo L, Gyaltsen P, Hudes M. Nutritional and health status of Tibetan children living at high altitudes. N Engl J Med. 2001 Feb 1;344(5):341-7. doi: 10.1056/NEJM200102013440504. PMID 11172165
- [Background] Utiger RD. Kashin-Beck disease--expanding the spectrum of iodine-deficiency disorders. N Engl J Med. 1998 Oct 15;339(16):1156-8. doi: 10.1056/NEJM199810153391611. No abstract available. PMID 9770565
- [Background] Chanoine JP. Selenium and thyroid function in infants, children and adolescents. Biofactors. 2003;19(3-4):137-43. doi: 10.1002/biof.5520190306. PMID 14757964
- [Background] Molecular Biology of selenium with its implications for metabolism. Raymond F. Burke, Division of Gastroenterology, division of Medicine and center in molecular toxicology, Vanderbilt University school of medicine, Nashville, Tenn 37232, USA